CLINICAL TRIAL: NCT01510535
Title: An Double-blind, Active-controlled, Parallel-group, Randomized, Multi-center Study to Compare Efficacy and Safety of LBSA0103 Once Versus Hyruan Plus Injection Once Weekly for 3weeks in the Treatment of Patients With Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of LBSA0103 Versus Hyruan Plus Injection in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-HACL010
Record Dates: First submitted 2012-01-06; First posted 2012-01-16 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoartritis; Knee; LBSA0103; Hyruan Plus Inj.
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo and then LBSA0103 (Experimental): The experimental group receive once weekly for 2 weeks intraarticular injections of Placebo(saline). And then, they receive once intraarticular injections of LBSA0103 into the target knee.
  Interventions: Drug: Placebo; Drug: LBSA0103
- Hyruan Plus (Active Comparator): The control group received once weekly for 3 weeks intraarticular injections of Hyruan Plus Inj. into the target knee.
  Interventions: Drug: Hyruan Plus

INTERVENTIONS:
Drug: Placebo — First 2 weeks Placebo(2ml) once weekly in experimental group
  Arms: Placebo and then LBSA0103
Drug: Hyruan Plus — Hyruan Plus Inj. (2ml)once weekly for 3 weeks in control group
  Arms: Hyruan Plus
Drug: LBSA0103 — at third week LBSA0103(60mg) once in experimental group
  Arms: Placebo and then LBSA0103

SUMMARY:
The purpose of this study is to compare efficacy and safety of intra-articular LBSA0103 once versus intra-articular hyaluronic acid injections (Hyruan Plus Injection) once weekly for 3 weeks in the treatment of patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years of age
* Kellgren & Lawrence grade I-III
* If there is more than one knee having a weight bearing pain of at least 40mm evaluated by 100mm VAS
* Be willing to discontinue all nonsteroidal anti-inflammatory drugs(NSAIDs), analgesics, condroichin sulfate/glucosamine or physical therapy for the duration of the study

Exclusion Criteria:

* Body mass index > 32
* Have rheumarthritis
* Patients who have a weight-bearing pain of less than 40mm on both knees when measured by 100mm-VAS
* Have Sudek's atrophy, Paget's disease, Spinal disc herniation
* Kellgren & Lawrence Grade IV

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Weight-bearing pain | 12 weeks after the last injection
  using 100mm-VAS

SECONDARY OUTCOMES:
Weight-bearing pain | 1,6 weeks after the last injection
  using 100mm-VAS
WOMAC-likert assessment | 1,6,12 weeks after the last injection
  Pain, Function, Stiffness, Total score
Patient Global Assessment | 1,6,12 weeks after the last injection
  using 100mm-VAS
Investigator Global Assessment | 1,6,12 weeks after the last injection
  using 100mm-VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Jongno-gu, Seoul, South Korea

REFERENCES:
- [Derived] Ha CW, Park YB, Choi CH, Kyung HS, Lee JH, Yoo JD, Yoo JH, Choi CH, Kim CW, Kim HC, Oh KJ, Bin SI, Lee MC. Efficacy and safety of single injection of cross-linked sodium hyaluronate vs. three injections of high molecular weight sodium hyaluronate for osteoarthritis of the knee: a double-blind, randomized, multi-center, non-inferiority study. BMC Musculoskelet Disord. 2017 May 26;18(1):223. doi: 10.1186/s12891-017-1591-4. PMID 28549436